CLINICAL TRIAL: NCT02312115
Title: DRAFFT Trial: Delayed Renal Allograft Function and Furosemide Treatment: A Randomized Prospective Double-blinded Placebo-controlled Clinical Pilot Trial
Brief Title: Delayed Renal Allograft Function and Furosemide Treatment
Acronym: DRAFFT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5140378
Record Dates: First submitted 2014-11-25; First posted 2014-12-09 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Delayed Graft Function
Keywords: Renal transplant; Kidney transplant; DGF
MeSH Terms: conditions — Delayed Graft Function | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide (Active Comparator): Patients assigned to the furosemide infusion group will receive furosemide infusions, as outlined in figure 2. This has been adapted from Ostermann et al. (2007) and the SPARK study protocol (Bagshaw et al. 2010). Furosemide will be prepared in bags that contain 1000 mg of furosemide per 250 mL of saline reaching a concentration of 4 mg/mL. All medication and placebo bags will have no identifiers that show what type of drug is being administered, for blinding purposes. Medication and placebo bags will have randomly generated study identifier numbers. The protocol in figure 2 will be followed to achieve a total urine output of 1mL/kg/h. The furosemide infusion rate will not exceed 4mg/min IV as this is the maximum set by the manufacturer.
  Interventions: Drug: Furosemide
- Saline (Placebo Comparator): All patients assigned to the saline group will receive saline that is equal in volume as compared to the treatment group. The amount of saline given to the patients in the placebo arm is so small that its effect on these patients is negligible. All other aspects of care for the enrolled patient will be managed per primary team and any consultants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Furosemide — Diuretic
  Other Names: Lasix
  Arms: Furosemide
Drug: Placebo — Saline
  Other Names: Saline placebo
  Arms: Saline

SUMMARY:
This study will be a randomized prospective double-blind placebo-controlled clinical pilot trial. This will be a single center project that will take place at Loma Linda University Medical Center. All adult kidney recipients will be informed of the study prior to operation. The Nephrology fellows or attending physicians will attempt to obtain informed consent from all eligible patients, pre-transplant. Those patients who consent will be screened post operation for enrollment. Patients who do not meet all eligibility criteria and/or who meet some exclusion criteria will be deemed ineligible for the trial, and will be excluded. The Nephrology and Transplant teams will be blinded of patient assignment and only the pharmacy will know the patient's assignment.

DETAILED DESCRIPTION:
1. Background/ Rationale Kidney Transplantation is a lifesaving modality in patients with end-stage renal disease (ESRD), and the numbers of transplants have been skyrocketing since the first successful trials. In 2013 alone, there were over 18,000 kidney transplants done in the United States of America. Of those, 11,161 were from a deceased donor (NKUDIC 2011, One Legacy 2014, USRDS 2013). One common complication of renal transplants is Delayed Graft Function (DGF). DGF is a serious complication, which is best defined as the need for renal replacement therapy, such as dialysis, within the first week after renal transplant (Mallon et al. 2013). DGF greatly increases the risk of acute and chronic transplant rejection, which decreases patient survival and quality of life, for those patients who do survive (Perico et al. 2004, Weber et al. 2014). Additionally, the rate of DGF is highest in patients who have received deceased donor transplants (One Legacy 2014). Therefore, it is crucial to the well-being of this large population to reduce the incidence of DGF. Our approach is to investigate current treatment modalities for patients post-deceased donor renal transplant, to understand how best to prevent DGF before it even starts. Currently, administration of loop diuretics such as furosemide is a common practice in order to prevent and treat oliguria in renal transplant patients. However, only animal models have been able to show a benefit in treating acute kidney injury (AKI), which occurs in the transplant kidney due to cold ischemia time, with furosemide. There is a lack of evidence that furosemide use leads to improved patient outcomes in patients with AKI (Nadeau-Fredette et al. 2013). Given that side effects of furosemide administration include ototoxicity, hypotension, electrolyte abnormalities, and hypersensitivity reactions, and the investigators hypothesize, may not significantly reduce the incidence of DGF from placebo, it is important to investigate if the benefits of furosemide administration truly outweigh the harms (Strom et al. 2003). The investigators intend to achieve this by way of a randomized, double-blinded, pilot clinical trial in adult oliguric patients, post-deceased donor renal transplant.
2. Objectives

I.Primary Objective:

i.To test the hypothesis that DGF rate is the same in adult oliguric post-deceased donor renal transplant patients administered furosemide vs. placebo.

II.Secondary Objectives:

i.To compare the following within the two treatment groups:

* 30-day, 90-day and 12-month creatinine levels and estimated glomerular filtration rate (eGFR)
* The need for RRT (Hemodialysis or Peritoneal dialysis) 30 days, 90 days and 12 months post-transplant
* The time from transplant to DGF development
* The incidence of DGF
* The incidence of primary graft non-function
* Overall hospital length of stay
* The KDPI score in relation to primary graft non-function

ii. To quantify the association between furosemide administration and relevant patient centered outcomes, such as hospital length of stay and acquired complications, in order to decrease patient morbidity and mortality.

c. Study Outline

All patients that have been admitted for a deceased donor kidney transplant will be seen by the Nephrology service for pre-transplant evaluation. The Nephrology Fellow/Attending physician will go over a checklist that determines if the patient will be eligible for the study and will obtain the informed consent if the patient is eligible. Informed consent will be obtained from all eligible patients. All eligible patients' urine output will be monitored as soon as they return to the unit from the operating room. If the patient remains oliguric or anuric for 6 hours, the bedside nurse will alert the on-call study coordinator for randomization and enrollment per protocol.

Study Intervention Patients assigned to the furosemide infusion group will receive furosemide infusions, as outlined in figure 2. This has been adapted from Ostermann et al. (2007) and the SPARK study protocol (Bagshaw et al. 2010).

Furosemide will be prepared in bags that contain 1000 mg of furosemide per 250 mL of saline reaching a concentration of 4 mg/mL. All medication and placebo bags will have no identifiers that show what type of drug is being administered, for blinding purposes. Medication and placebo bags will have randomly generated study identifier numbers. The protocol in figure 2 will be followed to achieve a total urine output of 1mL/kg/h. The furosemide infusion rate will not exceed 4mg/min IV as this is the maximum set by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with ESRD who has been on RRT (Hemodialysis or Peritoneal dialysis)
* Recipient of deceased donor kidney transplant
* Urine output less than 0.5 mL/kg/h before transplant
* Patient consents to the study
* Patient is not allergic to furosemide or sulfa
* English or Spanish speaking patient
* Patient is oliguric (urine output less than 0.5mL/kg/h, as per AKIN criteria) or anuric (urine output less than 10 mL in 6 hours post-transplant or 2 mL/h) in the first 6 hours post kidney transplant

Exclusion Criteria:

* Recipients of a living donor kidney transplant
* Patients who do not consent for the study
* Patients age <18 years
* Patients who are allergic to furosemide or sulfa containing medications
* Non-oliguric patients
* Patients who require immediate dialysis within 6 hours of the transplant (before enrollment)
* Patients with renal ischemia due to vascular compromise that has been confirmed with Doppler Ultrasound right after transplant as per standard of care
* Patients who return to the operating room due to complications within 24 hours
* Simultaneous multi-organ transplant recipients
* Hypotensive patients with BP <90/60 or MAP <60 mmHg
* Patients who are on vasopressors at any time during study period
* Non-English or Spanish speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The percent of participants receiving a deceased donor kidney that develop Delayed Graft Function (DGF), defined as the need to undergo Renal Replacement Therapy (RRT) within the first seven days after renal transplant. | 7 Days

SECONDARY OUTCOMES:
30-day, 90-day and 12-month creatinine levels and estimated Glomerular Filtration Rate (eGFR) | 30 days, 90 days and 12 months post-transplant
The need for Renal Replacement Therapy (RRT) 30 days, 90 days and 12 months post-transplant | 30 days, 90 days and 12 months post-transplant
The time from transplant to Delayed Graft Function (DGF) development | 24 hours
The incidence of Delayed Graft Function (DGF) | 24 Hours
The incidence of primary graft non-function | 12 months
Overall hospital length of stay | 30 days
The Kidney Profile Donor Index (KDPI) score in relation to primary graft non-function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Abdipour, MD, Principal Investigator — Attending Nephrologist, Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No